CLINICAL TRIAL: NCT00304265
Title: Reactogenicity of Acellular Pertussis Vaccine Booster in Adolescents Who Have Received 5 Prior Doses of BIKEN Acellular Pertussis Vaccine in Combination With Diphtheria and Tetanus Toxoids (TRIPEDIA®) or Who Have Received Primary Vaccination With 3 Doses of Whole-Cell Pertussis Vaccine, Plus at Least 1 Pertussis Booster Vaccination
Brief Title: Post-marketing Evaluation of Reactions Following Receipt of Recommended Adolescent Pertussis Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRI05
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Results first posted 2011-04-07 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Pertussis; Diphtheria; Tetanus; Poliomyelitis
Keywords: Pertussis,; Diphtheria,; Tetanus,; Poliomyelitis
MeSH Terms: conditions — Whooping Cough; Diphtheria; Tetanus; Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6th Dose Pertussis Vaccine Group (Experimental): Participants received 6th dose of pertussis vaccine
  Interventions: Biological: COVAXIS™: Tetanus, diphtheria, acellular 5-component pertussis, or + inactivated poliovirus vaccine (REPEVAX®)
- 5th Dose Pertussis Vaccine Group (Experimental): Participants received 5th dose of pertussis vaccine
  Interventions: Biological: COVAXIS™: Tetanus, diphtheria, acellular 5-component pertussis, or + inactivated poliovirus vaccine (REPEVAX®)

INTERVENTIONS:
Biological: COVAXIS™: Tetanus, diphtheria, acellular 5-component pertussis, or + inactivated poliovirus vaccine (REPEVAX®) — 0.5 mL, Intramuscular
  Other Names: REPEVAX®; COVAXIS™; IPV Merieux™

SUMMARY:
Post-marketing evaluation of reactions following receipt of recommended adolescent pertussis vaccine among persons with prior vaccination with acellular vs whole-cell pertussis vaccine.

To describe and characterize adverse events occurring after vaccination with REPEVAX® (Tdap-IPV: combination diphtheria, tetanus and acellular pertussis with inactivated poliomyelitis vaccine) or COVAXIS® (Tdap: combination diphtheria, tetanus and acellular pertussis) vaccine among two groups: Group 1 - adolescents 10-14 years of age who participated in study 371-03/01 (and thus received a 5th dose of TRIPEDIA® vaccine) and Group 2 - controls 10-14 years of age who were vaccinated with at least three doses of a whole-cell pertussis vaccine in infancy plus at least one subsequent dose of pertussis vaccine in their 2nd through 7th year of life.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive REPEVAX® or COVAXIS® vaccine, in accord with German recommendations for a booster dose of acellular pertussis vaccine at 9-17 years of age.
* Signed and dated informed consent or assent form (as applicable) that is obtained prior to the first study intervention.
* Judged to be in good health on the basis of reported medical history and history-directed physical examination.
* Plans to remain in the study area for the length of the trial.
* The participant and a parent or legal guardian can read, write, and understand the documents and all are mentally competent to give assent and consent.
* If female, not known or suspected to be pregnant at the time of enrollment into the study and is not planning pregnancy during participation in this trial.
* Either prior participation in study 371-03/01 (Group 1 - 6th Dose Pertussis Vaccine Group) or a documented history of 3 doses of tetanus, diphtheria and whole-cell pertussis vaccine in infancy plus at least one subsequent dose of pertussis vaccine in their 2nd through 7th year of life (Group 2 - 5th Dose Pertussis Vaccine Group).
* Has access to a telephone.
* Oral temperature < 38.0ºC.

Exclusion Criteria:

* Pregnancy or nursing a child
* Known or suspected primary or acquired disease of the immune system (conditions suspected of having an immunologic component such as autoimmune diseases [e.g. rheumatoid arthritis or inflammatory bowel disease] will not be excluded unless they meet exclusion criterion 3 or 5).
* Malignancy, allergy immunotherapy, or receiving immunosuppressive therapy (participants who are taking topical and inhaled steroids could be included in the study as would participants on a "short course" of oral steroids, -<7 days, as long as there are not two courses within the previous two weeks prior to vaccination).
* Receipt of any pertussis, diphtheria or tetanus-containing vaccines within the past 3 years.
* Any unstable significant underlying chronic disease, including (but not limited to) malignancy, cardiopulmonary disease, renal, endocrinologic, hematologic or hepatic dysfunction.
* Known impairment of neurologic function or currently active seizure disorder or currently requiring medication for seizures.
* Personal history of physician-diagnosed or laboratory-confirmed pertussis disease within the last 2 years.
* Receipt of blood products or immunoglobulin within the previous 3 months.
* Known or suspected allergy to any of the vaccines or vaccine components intended for use in the study.
* Daily use of non-steroidal anti-inflammatory drugs.
* Receipt of any vaccine or investigational product within the 30 days prior to enrollment, or planning to receive another vaccine within 28 days after receiving study vaccine.
* Chemical dependency (e.g. alcoholism or intravenous drug use but not including nicotine or caffeine), based on investigator judgment.
* Known or suspected acute infectious respiratory illness at the time of vaccination with active symptoms and signs including one or more of the following: rhinorrhea, new cough, pharyngitis, respiratory problems (e.g. wheezing, shortness of breath).
* Any condition which, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* History of immediate anaphylaxis, encephalopathy within 7 days, or seizure within 3 days of receiving diphtheria, tetanus, or pertussis vaccine.
* Planned participation in another interventional clinical trial during the present trial period (participation in a related study to evaluate immune responses to this study's vaccination is permitted).
* Thrombocytopenia or bleeding disorder that would pose a contraindication to an intramuscular (IM) vaccination.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 215 (Actual)
Dates: Start 2006-03; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (16):
- Germany (16):
  - Munich, Lindwurmstrasse 4
  - Bielefeld
  - Detmold
  - Donzdorf
  - Grafing
  - Heilbronn
  - Lauffen am Neckar
  - Marbach
  - Marktoberdorf
  - Munich
  - Schwandorf in Bayern
  - Schwäbisch Hall
  - Schwieberdingen
  - Stuttgart
  - Süßen
  - Veitshöchheim

REFERENCES:
- [Result] Liese JG, Rieber N, Malzer T, Ocak M, Johnson DR, Decker MD; Munich Vaccine Study Group. Reactogenicity of tetanus, diphtheria, 5-component acellular pertussis vaccine administered as a sixth consecutive acellular pertussis vaccine dose to adolescents. Pediatr Infect Dis J. 2010 Dec;29(12):1067-71. doi: 10.1097/INF.0b013e3181ea5866. PMID 20616762
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February 2006 to July 2006 at 17 clinical sites in Germany.
Pre-assignment Details: A total of 214 participants who met the inclusion and exclusion criteria were enrolled and vaccinated. One over aged participant was also vaccinated and included in the safety analysis.
Groups:
- 6th Dose Pertussis Vaccine Group: Participants who had received 5 doses of BIKEN acellular pertussis vaccine in Study 371-03/01 received REPEVAX® (Tdap-IPV: combination diphtheria, tetanus and acellular pertussis with inactivated poliomyelitis vaccine) or COVAXIS® (Tdap: combination diphtheria, tetanus and acellular pertussis) vaccine as a 6th (booster) dose as adolescents.
- 5th Dose Pertussis Vaccine Group: Participants who had received at least 3 doses of whole-cell pertussis vaccine during infant immunization and at least 1 subsequent booster vaccination in the 2nd to 7th years of life received either REPEVAX® (Tdap-IPV: combination diphtheria, tetanus and acellular pertussis with inactivated poliomyelitis vaccine) or COVAXIS® (Tdap: combination diphtheria, tetanus and acellular pertussis) vaccine as a 5th (booster) dose as adolescents.
Period: Overall Study
Arm/Group | 6th Dose Pertussis Vaccine Group | 5th Dose Pertussis Vaccine Group
Started | 117 | 98
Completed | 117 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6th Dose Pertussis Vaccine Group | 5th Dose Pertussis Vaccine Group | Total
Number analyzed (Participants) | 117 | 98 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 117 | 98 | 215
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 12.3 (0) [11 to 13] | 12.6 (0) [10 to 16] | 12.4 (0) [10 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 37 | 92
  Male | 62 | 61 | 123
Region of Enrollment [Number; unit: Participants]
  Germany | 117 | 98 | 215

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting a Solicited Local or Systemic Reaction Post-Vaccination With Either REPEVAX® or COVAXIS® Vaccine
Description: Solicited injection site reactions: Pain, Erythema, Swelling, and Arm circumference.
  Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia.
Time Frame: Days 0 to 14 Post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | 6th Dose Pertussis Vaccine Group | 5th Dose Pertussis Vaccine Group
Number analyzed (Participants) | 117 | 97
Participants
  Any Local Reactions After Vaccination | 89 | 87
  Any Pain | 85 | 87
  Grade 3 Pain (Incapacitating) | 7 | 8
  Any Erythema | 19 | 27
  Grade 3 Erythema (> 5.0 cm) | 10 | 10
  Any Swelling | 24 | 17
  Grade 3 Swelling (> 5.0 cm) | 6 | 8
  Any Increase in Arm Circumference | 8 | 11
  Grade 3 Increase in Arm Circumference (> 5.0 cm) | 0 | 0
  Any Systemic Reactions After Vaccination | 85 | 84
  Fever | 5 | 15
  Any Headache | 40 | 50
  Grade 3 Headache (Prevents Daily Activities) | 4 | 5
  Any Malaise | 40 | 44
  Grade 3 Malaise (Prevents Daily Activities) | 2 | 2
  Any Myalgia | 69 | 73
  Grade 3 Myalgia (Prevents Daily Activity) | 5 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 28 days post-vaccination.
Arm/Group | 6th Dose Pertussis Vaccine Group | 5th Dose Pertussis Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/117 | 0/98
Other Adverse Events (participants affected / at risk) | 89/117 | 87/97
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6th Dose Pertussis Vaccine Group (N=117) | 5th Dose Pertussis Vaccine Group (N=97)
Injection site pain (General disorders) | 89 | 87
Injection site erythema (General disorders) | 19 | 27
Injection site swelling (General disorders) | 24 | 17
Headache (Nervous system disorders) | 40 | 50
Malaise (General disorders) | 40 | 44
Myalgia (Musculoskeletal and connective tissue disorders) | 69 | 73
Pyrexia (General disorders) | 5 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.